CLINICAL TRIAL: NCT07058870
Title: Unravelling The Optimisation And Consolidation Of Motor Skills In People With Multiple Sclerosis With Mild to Moderate Gait Impairment Via High Intensity Task Oriented Circuit Training: A Feasibility Study
Brief Title: Unravelling The Optimisation And Consolidation Of Motor Skills In People With Multiple Sclerosis With Mild to Moderate Gait Impairment: A Feasibility Study
Acronym: UNLOCK MS MGI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, PhD, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLOCK_MS_MGI_HITOCT
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: high intensity training; multiple sclerosis; motor learning; mild to moderate multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: High Intensity Task Oriented Circuit Training + Telerehabilitation (Experimental): Participants will receive 10 sessions (one hour each, three times a week) including structured exercise stations targeting key motor skills such as walking, walking adaptability, stepping and supine to stand transition.
  Afterwards, participants will engage in 36 sessions (30 minutes each, three times a week) of asynchronous telerehabilitation targeting supine to stand transition, stepping and walking.
  Interventions: Behavioral: High Intensity Task Oriented Circuit Training + Telerehabilitation

INTERVENTIONS:
Behavioral: High Intensity Task Oriented Circuit Training + Telerehabilitation — Participants will receive 10 sessions of high-intensity, task-oriented circuit training, three times a week. Each session will last 60 minutes, with minutes of active training. Each session will include three rounds, each lasting 55 minutes. During each round, participants will rotate between stations working for four minutes at each station, followed by three minutes of rest. The stations will focus on key motor skills, including supine to stand transitions, walking speed and functional capacity, walking adaptability and stepping. After in-hospital treatment participants will receive 36 sessions of asynchronous telerehabilitation, three times a week for 12 weeks. This intervention will be supported by low-cost, off-the-shelf technology for treatment delivery and monitoring.

SUMMARY:
The goal of this feasibility study is to test the safety and effectiveness of an high-intensity task oriented circuit training program, followed by three months of telerehabilitation in people with mild to moderate Multiple Sclerosis (MS). The main questions it aims to answer are:

* Can high-intensity task oriented circuit training improve gait and balance functional capacity?
* Can telerehabilitation mantain the benefits in gait and balance gained via circuit training for a six month period?

Participants will:

* Complete 10 session ( one hour each, three times a week) of high-intensity task oriented circuit training administered in a hospital setting. The training will target key motor skills such as walking, stepping, supine to stand transitions and general mobility.
* Engage in 3 months of asynchronous telerehabilitation (without physiotherapist supervision)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary progressive multiple sclerosis according to the McDonald criteria.
* Mini-Mental State Examination (MMSE) score > 24.
* Expanded Disability Status Scale (EDSS) score ≤ 6.

Exclusion Criteria:

* Presence of other psychiatric or neurological disorders.
* Cardiopulmonary, renal, or liver diseases.
* Pregnancy.
* Modifications in drug treatment within the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Balance | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The change in balance will be assessed using the Fullerton Advanced Balance Scale

SECONDARY OUTCOMES:
Change in mobility, balance, walking ability, and fall risk | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Mobility, balance, walking ability, and fall risk will be assessed through Timed Up and Go Test
Change in Dual task Cost | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Dual Task Cost will be assessed by the difference between Timed Up and Go and Dual Task Timed Up and Go
Change in quantitative mobility and leg function performance | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Leg function performance and quantitative mobility assessed through Timed 25 Foot Walk
Change in auditory information processing speed and flexibility | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Paced Auditory Serial Addition Test will be used to assess auditory information processing speed and flexibility
Change in Walking Speed | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  10 Meters Walking Test will be used to assess the change in walking speed
Change in ability to modify balance while walking in the presence of external demands | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The extended version of the Dynamic Gait Index will be used to assess ability to modify balance while walking in the presence of external demands
Change in dynamic balance during an activity requiring weight-shift and movement while in single-leg stance | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Step Test will be used to assess the change in dynamic balance during an activity requiring weight-shift and movement while in single-leg stance
Change in ability to transition from a supine positon to a standing position. | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The Supine To Stand Test will be used to assess the ability to transition from a supine positon to a standing position.
Change in functional lower extremity strength | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Five Times Sit to Stand will be used to assess functional lower extremity strength
Change in Walking capacity | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Walking capacity will be assessed through the 6 Minute Walking Test
Change in Subjective Trait Fatigue | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Change in subjective trait fatigue will be assessed through Modified Fatigue Impact Scale
Change in impacts of multiple sclerosis in people' lifes | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The impact of multiple sclerosis in people' lifes will be assessed through Multiple Sclerosis Impact Scale 29.
Change in balance confidence | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Change in balance confidence will be assessed through Activity-Specific Balance Confidence Scale.
Change in perceieved impact of MS on the individual's walking ability. | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The 12-item Multiple Sclerosis Walking Scale (MSWS-12) will be used to measure of the impact of MS on the individual's walking ability.
Change in Walking Fatigability | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The Distance Walking Index will be used to assess the Change in Walking Fatigability

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrara University Hospital, Ferrara, FE, Italy